CLINICAL TRIAL: NCT04201054
Title: Generation of Biological Samples Positive to Fluconazole for Anti-Doping Control
Acronym: FLUC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMIMFTCL/FLUC
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers
Keywords: Fluconazole; Anti-doping control; Athletic performance
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluconazole (Experimental): Subjects receive a single-dose treatment.Urine samples will be collected after administration (4 fractions: 0-12, 12-24, 24-48, 48-72 hours post-administration).
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — 50 mg of fluconazole administered orally in a single dose.

SUMMARY:
Background:

Androgens are used for doping purpose because they can increase muscle mass and strength. These drugs are included in the list of prohibited substances of the World Anti-Doping Agency (WADA). The prohibition of its use has given rise to a great variety of strategies, including indirect androgenic doping (increasing endogenous testosterone production) or masking of exogenous testosterone administration.

Fluconazole is an imidazole antifungal that inhibits certain cytochrome P-450 dependent enzymes participating in the synthesis of steroid hormones. Concomitant fraudulent administration of testosterone and fluconazole may cause lower steroid concentrations in urine, leading to false negatives in the doping control. Thus, fluconazole may be used in athletes to mask exogenous steroid administration.

Hypothesis:

The oral administration of 12,5 mg of hydrochlorothiazide in healthy subjects allows generating detectable concentrations of the drug in urine. Positive urine samples will enable to identify analytical strategies for doping control.

Objectives:

Primary objective: To measure the concentrations of fluconazole in urine for anti-doping control samples.

Secondary objectives: To identify fluconazole metabolites in urine. To explore the time window in which the drug or its metabolites can be detected in urine after administration. To assess safety and tolerability of the drug used.

Methods:

Phase I, open, non-randomized clinical trial, with a treatment condition (fluconazole) administered in a single oral dose to 2 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers aged between 18 and 45 years.
* Able to understand and accept the trial procedures and able to sign an informed consent.
* History and physical examination that demonstrate not presenting organic or psychiatric disorders.
* ECG, blood and urine tests performed at screening should be within normal limits. Minor or punctual variations of these limits of normality are admitted if, in the opinion of the Principal Investigator, they have no clinical significance, do not pose a risk to the subject and do not interfere with the evaluation of the product in study. These variations and their nonrelevance will be justified in writing specifically.
* Body mass index (weight/size^2) between 19 and 25 kg/m2. Subjects with BMI between 25-27 kg/m2 may be included at the discretion of the Principal Investigator.

Exclusion Criteria:

* Failure to meet the inclusion criteria.
* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active substance or any of the excipients.
* History of serious adverse reactions to other medications.
* Subjects with contraindications to treatment with the study drug (according to Summary of Product Characteristics).
* Background or clinical evidence of psychiatric disorders, alcoholism, regular consumption of psychoactive drugs, drug abuse or addiction to other substances (except for nicotine).
* Smokers of more than 20 cigarettes/day in the 3 months prior to the start of the study.
* Having participated in another clinical trial with medication in the three months prior to the start of the study.
* Having donated blood in the 2 months prior to the start of the study.
* Having suffered an organic disease or major surgery in the 6 months prior to the start of the study.
* Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological, dermatological or other acute or chronic diseases that, in the opinion of the Principal Investigator or the collaborators designated by him, may pose a risk to the subjects, may interfere with the objectives of the study or may alter the pharmacokinetics of the drug. Especially in case of seizures or history of epilepsy.
* Having taken medication regularly in the month prior to the study sessions, with the exception of vitamins, herbal remedies or dietary supplements that, in the opinion of the Principal Investigator or the collaborators designated by him, do not pose a risk to the subjects and do not interfere with the objectives of the study. Treatment with single doses of symptomatic medication in the week prior to the study sessions will not be exclusive if it is assumed that medication has been completely eliminated on the day of the experimental session.
* Consumption of more than 40 g of alcohol per day.
* Consumers of more than 5 coffees, teas, cola drinks and/or other stimulant drinks (xanthines) per day in the 3 months prior to the start of the study.
* Being unable to understand the nature of the trial and the procedures requested to follow.
* Positive serology for hepatitis B, C or HIV.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Urine concentration of fluconazole | 0-12 hours post-administration
  Concentration of fluconazole in fraction-1 urine samples
Urine concentration of fluconazole | 12-24 hours post-administration
  Concentration of fluconazole in fraction-2 urine samples
Urine concentration of fluconazole | 24-48 hours post-administration
  Concentration of fluconazole in fraction-3 urine samples
Urine concentration of fluconazole | 48-72 hours post-administration
  Concentration of fluconazole in fraction-4 urine samples

SECONDARY OUTCOMES:
Urine concentration of fluconazole metabolites | 0-12 hours post-administration
  Concentration of fluconazole metabolites in fraction-1 urine samples
Urine concentration of fluconazole metabolites | 12-24 hours post-administration
  Concentration of fluconazole metabolites in fraction-2 urine samples
Urine concentration of fluconazole metabolites | 24-48 hours post-administration
  Concentration of fluconazole metabolites in fraction-3 urine samples
Urine concentration of fluconazole metabolites | 48-72 hours post-administration
  Concentration of fluconazole metabolites in fraction-4 urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Rafael de la Torre Fornell, Dr, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No